CLINICAL TRIAL: NCT05274438
Title: A Single-arm, Phase II Clinical Study of Imatinib Mesylate Combined With Toripalimab in the Treatment of Stage III Unresectable and Stage IV Melanoma Harbored With CKIT Mut
Brief Title: Imatinib and Toripalimab in Patients With Locally Advanced/Metastatic Melanoma Harbored With CKIT Mut
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO208
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS001+Imatinib Mesylate (Experimental): Imatinib: 400mg qd po. Toripalimab: 240mg q3w ivgtt. The longest cumulative use period of the two drugs was 2 years.
  Interventions: Drug: JS001+Imatinib mesylate

INTERVENTIONS:
Drug: JS001+Imatinib mesylate — This study consisted of two phases: the first phase was the dose exploration phase, and the second phase was the extension group. In phase I, 3 patients were enrolled, starting with imatinib monotherapy, 400mg qd, for 2 cycles (6 weeks), followed by imatinib 400mg qd combined with toripalimab 240mg q3w. If DLT was not observed, the original dose was extended to 37 patients in phase ii; If there was 1 DLT in the first stage, the number of patients in the first stage was extended to 6. If there was no DLT, the patients entered the extended stage. If ≥2 DLT cases occurred in the first phase, imatinib was reduced to 300mg QD and toripalimab 240mg q3W, and the "3+3" study was restarted. If DLT≤1 case, enter extended group (imatinib 300mg qd and toripalimab 240mg q3W); The longest cumulative use period of the two drugs was 2 years. When patients develop disease progression or develop intolerable toxicity, treatment is ended and follow-up for survival is entered.

SUMMARY:
It is a single-center, single-arm Phase II clinical study. This clinical trial aimed to evaluate the PFS of imatinib combined with toripalimab in stage III unresectable and stage IV melanoma with CKIT gene mutation.

DETAILED DESCRIPTION:
This study consisted of two phases: the first phase was the dose exploration phase, and the second phase was the extension group. In phase I, 3 patients were enrolled, starting with imatinib monotherapy, 400mg qd, for 2 cycles (6 weeks), followed by imatinib 400mg qd combined with toripalimab 240mg q3w. If DLT was not observed, the original dose was extended to 37 patients in phase ii; If there was 1 DLT in the first stage, the number of patients in the first stage was extended to 6. If there was no DLT, the patients entered the extended stage. If ≥2 DLT cases occurred in the first phase, imatinib was reduced to 300mg QD and toripalimab 240mg q3W, and the "3+3" study was restarted. If DLT≤1 case, enter extended group (imatinib 300mg qd and toripalimab 240mg q3W); The longest cumulative use period of the two drugs was 2 years. When patients develop disease progression or develop intolerable toxicity, treatment is ended and follow-up for survival is entered.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, no gender limitation;
2. Patients with recurrent, unresectable or metastatic melanoma confirmed by histopathology after surgery (stage III/IV);
3. With CKIT gene mutation;
4. Did not receive CKIT inhibitor or PD-1/PD-L1 mab treatment in late stage; Adjuvant therapy Patients who have received CKIT inhibitors or PD-1/PD-L1 mab should be discontinued for at least 6 months;
5. ECOG score is 0 or 1;
6. Expected survival ≥3 months;
7. The investigator assessed the presence of at least one measurable lesion that had not been irradiated according to RECIST 1.1;
8. No history of brain/meningeal metastasis;
9. The organ function level must meet the following requirements (7 days before the first administration of the study drug):

   Spinal cord: Neutrophil absolute count (ANC)≥1.5×109/L, platelet (PLT)≥ 100×109/L, and hemoglobin (HB)≥9g/dL(no blood transfusion or component blood was received within 14 days prior to test); Gallo liver: Serum total bilirubin (TBIL)≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5 times the upper limit of normal ( allows AST and ALT≤5 times the upper limit of normal if liver metastasis is present); serum creatinine ≤1.5 times the upper limit of normal value and endogenous creatinine clearance ≥50mL/min (Cockcroft-Gault formula); Accidence International standardized ratio (INR), activated partial thrombin time (aPTT)≤1.5 times the upper limit of normal value (only for patients not receiving anticoagulant therapy; Patients receiving anticoagulant therapy should keep the anticoagulant within the therapeutic range); Thyroid stimulating hormone (TSH)≤1×ULN (if abnormal, FT3 and FT4 levels should be investigated simultaneously; if FT3 and FT4 levels are normal, they can be included in the group) Isogenic urinary protein ≤1+, isogenic urinary protein & GT; 1+, urine protein should be collected for 24 hours, and the total amount should be less than or equal to 1 g; Unconsciously the heart functions normally, meaning normal or abnormal ECG has no clinical significance, while cardiac ultrasound shows left ventricular ejection fraction (LVEF) greater than 50%.
10. Serum pregnancy test results of women of childbearing age should be negative within 7 days before the first administration of the test drug; Men who are fertile or women who are at risk of becoming pregnant must use a highly effective method of contraception (e.g., oral contraceptives, intrauterine devices, abstinence of sex or barrier contraception combined with spermicide) throughout the trial and continue to use contraception for 180 days after completion of treatment;
11. Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

1. Advanced treatment with CKIT inhibitors or PD-1/PD-L1 mab; Adjuvant therapy received CKIT inhibitor or PD-1/PD-L1 mab, and the drug withdrawal was less than 6 months;
2. Associated with cerebral/meningeal metastasis;
3. Patients who participated in or are participating in clinical trials of other drugs/therapies within 4 weeks prior to the first administration of the study drug;
4. The study drug underwent/underwent major surgery or had not yet recovered from the side effects of the surgery, received live vaccination, immunotherapy, and received radiotherapy within 2 weeks before the first administration of the study drug;
5. The patient has any active autoimmune disease or a history of autoimmune disease (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism); Vitiligo that does not require systemic treatment may be included; Asthma with complete remission in childhood and without any intervention in adulthood could be included; Patients with asthma requiring medical intervention with bronchodilators were excluded);
6. The patient is on immunosuppressant, or systemic hormone therapy for immunosuppression purposes (dose > 10mg/ day of prednisone or other equivalent hormone) and continued to use within 2 weeks prior to enrollment;
7. A history of malignancies other than melanoma in the past 5 years, with the exception of cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early-stage prostate cancer and carcinoma in situ of the cervix;
8. Patients who had received hematopoietic stimulating factors, such as granulocyte colony stimulating factor (G-CSF) and erythropoietin, within 1 week before the first drug administration;
9. Positive HIV antibody or treponema pallidum antibody;
10. Patients with active hepatitis B or C:

    If HBsAg or HBcAb is positive, add test for HBV DNA(test result is higher than the upper limit of the normal range).

    If HCV antibody test result is positive, add test HCV RNA(test result is higher than normal value fan circumference upper limit);
11. Known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components; Known to be allergic to imatinib mesylate and any excipients;
12. Large pleural effusion, ascites and pericardial effusion accompanied by clinical symptoms and requiring symptomatic treatment;
13. History of active pulmonary disease (interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or active pulmonary tuberculosis;
14. Have any clinical problems beyond control, including but not limited to:

    Either a persistent or active (severe) infection; Hypoglycemic medication for poorly controlled hypertension (persistent blood pressure greater than 150/90 MMHG) Buying something to control diabetes poorly; Buying a ticket for heart disease (class III/IV congestive heart failure or heart block, as defined by the New York Cardiology Society); Anyway, something happened during the first six months before taking the drug: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina pectoris; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; Cerebrovascular accident, transient ischemic attack, cerebral embolism;
15. Any conditions of the patient that affect the ingestion of the drug by the subject, and any conditions that affect the in-body disposal of the drug (absorption, distribution, metabolism or excretion);
16. Abnormal coagulation (INR> 2.0, PT> 16s), have bleeding tendency or are receiving thrombolytic or anticoagulant therapy, and are allowed to use low-dose aspirin and low-molecular weight heparin prophylacically;
17. The group of the first 3 months there have been significant clinical significance of bleeding symptoms or have a definite bleeding tendency, such as daily cough/haemoptysis 2.5 ml and above, gastrointestinal bleeding, there is a risk of bleeding of esophageal gastric varices, hemorrhagic peptic ulcers, or patients with vasculitis, baseline period if defecate occult blood positive, to review, after review if still positive, the need for gastroscopy, If severe esophagogastric fundus varices were indicated by gastroscopy, they could not be enrolled in the group (except those who were excluded by gastroscopy within 3 months before enrollment).
18. Known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulopathy, thrombocytopenia, etc.);
19. Have undergone a stem cell or organ transplant;
20. Those who have a history of psychotropic drug abuse and cannot get rid of it or have a history of mental disorders;
21. The investigator identifies other severe, acute, or chronic medical conditions or laboratory abnormalities that may increase the risk associated with study participation or may interfere with the interpretation of study results;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  To evaluate progression-free survival (PFS) based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  To evaluate the overall response rate (ORR) based on RECIST 1.1 criteria.
Disease control rate (DCR) | 2 years
  To evaluate the disease control rate (DCR) based on RECIST 1.1 criteria.
Overall survival (OS) | 2 years
  To evaluate overall survival (OS) based on RECIST 1.1 criteria.
Safety(AE,SAE) | 2 years
  To evaluate safety(AE,SAE) of imatinib mesylate combined with terriprizumab in patients with stage III unresectable and stage IV melanoma with CKIT gene mutation.

CONTACTS AND LOCATIONS:
Overall Officials: jun Guo, Diretcor, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo J, Si L, Kong Y, Flaherty KT, Xu X, Zhu Y, Corless CL, Li L, Li H, Sheng X, Cui C, Chi Z, Li S, Han M, Mao L, Lin X, Du N, Zhang X, Li J, Wang B, Qin S. Phase II, open-label, single-arm trial of imatinib mesylate in patients with metastatic melanoma harboring c-Kit mutation or amplification. J Clin Oncol. 2011 Jul 20;29(21):2904-9. doi: 10.1200/JCO.2010.33.9275. Epub 2011 Jun 20. PMID 21690468